CLINICAL TRIAL: NCT06745141
Title: Oral Health Intervention Study in Patients with Myocardial Infarction and Periodontal Disease: a Simulated RCT Trial
Brief Title: Myocardial Infarction and Periodontitis: Periodontal Health Intervention.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, professor of medicine, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCS-MIP-PHI
Record Dates: First submitted 2024-12-10; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Acute Myocardial Infarction (AMI); Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: This study employs a simulated randomized controlled trial (RCT) design to evaluate the effects of periodontal health interventions on patients with myocardial infarction (MI) complicated by periodontitis.
  The study mimics the framework of a traditional randomized controlled trial but does not involve formal randomization of participants.
  Participants are allocated into intervention and control groups in a structured manner to minimize bias, ensuring comparability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Periodontal Health Intervention Group (Experimental): Participants in this arm will receive comprehensive periodontal health interventions, including:
  1. Full periodontal evaluation using dental mirrors and probes (assessing visible plaque, probing depth, bleeding on probing, and attachment loss).
  2. Supragingival scaling, root planing, and professional plaque removal.
  3. Temporary restoration of carious lesions and extraction of root remnants, as needed.
  4. Personalized oral hygiene instruction, including the use of multi-tufted brushes, toothpaste, floss, and interdental brushes.
  Interventions: Procedure: Periodontal surgery
- Standard Care Group (No Intervention): Participants in this arm will receive standard care without specific periodontal interventions. This includes routine medical management for myocardial infarction, as per standard clinical guidelines, without structured periodontal treatment.

INTERVENTIONS:
Procedure: Periodontal surgery — In the intervention group, patients underwent a comprehensive periodontal evaluation conducted by periodontists at a dental clinic. All permanent teeth, except for third molars, were assessed using dental mirrors and periodontal probes. Each tooth was examined at four sites (vestibular, distal, lingual, and mesial) to evaluate visible plaque, probing depth, probing bleeding, and attachment loss.
  During the first treatment session, patients were provided with information about periodontal disease, emphasizing the importance of controlling supragingival bacterial biofilms for successful treatment. Plaque-retentive factors (calculus) were removed. Temporary materials were used to restore carious lesions, root remnants were extracted, and maladaptive restorations were adjusted. Supragingival calculus was removed using periodontal scalers, followed by cleaning with a rubber cup, prophylaxis paste, dental floss, and/or interdental brushes. No prophylactic antibiotics were used prior to the
  Arms: Periodontal Health Intervention Group

SUMMARY:
The aim of this study is to establish a shared database of acute myocardial infarction patients with periodontitis, to clarify the clinical benefits of periodontitis intervention on acute myocardial infarction patients through simulated RCT study, and to establish a high-level database of acute myocardial infarction patients with periodontitis, so as to promote the application of oral health intervention in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 1)Patients diagnosed with ST-segment elevation myocardial infarction (STEMI). 2)Patients with severe periodontal disease, defined as:

  * 5 teeth with clinical attachment loss (CAL) ≥ 4 mm.

    * Subgingival probing depth (PD) ≥ 6 mm. ③≥ 8 teeth with gingival bleeding on probing (BOP). 3）Age ≥30 years. 4）Written informed consent provided.

Exclusion Criteria:

* 1) under 30 years old; 2) HIV positive, chronic inflammation, tumor disease, drug dependence, use of anticonvulsants, use of immunosuppressive agents, pregnancy, and lactation; 3) significant tooth loss (number of remaining teeth < 8); 4) long hospital stay (>10 days), new myocardial infarction before randomization, and stent thrombosis; 5) Refusal to sign informed consent.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in ejection fraction | From enrollment to the end of treatment at 6 months
  The ejection fraction (EF) changed by 10% half a year after surgery

SECONDARY OUTCOMES:
Cardiovascular death and MACE events were recorded | From enrollment to the end of treatment at 6 months, a maximum of 12 months.
level of proBNP | From enrollment to the end of treatment at 6 months
  The outcome will be assessed by measuring the level of plasma N-terminal pro-B-type natriuretic peptide (NT-proBNP), a biomarker reflecting cardiac stress and heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China